CLINICAL TRIAL: NCT01422408
Title: Phase II Study of the Effect of the Topical Corticosteroid Fluocinonide in Patients on Endocrine Therapy for Either Breast Cancer or an Increased Risk for Breast Cancer With Symptoms of Vaginal Dryness and Dyspareunia
Brief Title: Fluocinonide Cream in Treating Symptoms of Vaginal Dryness and Painful Sexual Intercourse In Patients With Breast Cancer Undergoing Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kathleen Kemmer, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00007265; NCI-2011-01234 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CPC-11028-L (Other: OHSU Knight Cancer Institute); 7265 (Other: OHSU Knight Cancer Institute); P30CA69533OD (Other Grant/Funding Number: National Cancer Institute); P30CA069533 (NIH)
Record Dates: First submitted 2011-08-22; First posted 2011-08-24 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-07

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluocinonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (fluocinonide cream) (Experimental): Patients apply topical fluocinonide cream BID in weeks 1-2 and QD in weeks 3-4.
  Interventions: Drug: Fluocinonide Cream; Procedure: Management of Therapy Complications; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Fluocinonide Cream — Given topically
  Other Names: fluocinonide; Lidex; Vanos
Procedure: Management of Therapy Complications — Receive fluocinonide cream
  Other Names: complications of therapy, management of
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well giving fluocinonide cream works in treating symptoms of vaginal dryness and painful sexual intercourse in patients with breast cancer undergoing hormone therapy. Fluocinonide cream may prevent or lessen vaginal dryness and painful sexual intercourse in patients undergoing hormone therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the decrease in symptoms of vaginal dryness and dyspareunia with the use of fluocinonide 0.05% cream in breast cancer subjects and subjects at increased risk for breast cancer on endocrine therapy. Estimates of decrease will be obtained utilizing patient survey instruments.

SECONDARY OBJECTIVES:

I. To estimate the decrease in symptoms of vaginal itching and the total vaginal index score with the use of fluocinonide 0.05% cream in breast cancer subjects and subjects at increased risk for breast cancer on endocrine therapy. Estimates of decrease will be obtained utilizing patient survey instruments.

II. To explore toxicities reported by subjects using fluocinonide 0.05% cream via vaginal application.

III. To explore correlation between subject reported compliance, as well as compliance via measurement of the amount of fluocinonide 0.05% cream used, and response rates with the use of fluocinonide 0.05% cream.

IV. To explore the correlations between patient characteristics and response rates with the use of fluocinonide 0.05% cream.

OUTLINE:

Patients apply topical fluocinonide cream twice daily (BID) in weeks 1-2 and once daily (QD) in weeks 3-4.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (both pre-menopausal and post-menopausal women are eligible) and with a history of breast cancer or with an increased risk for breast cancer on current treatment with tamoxifen or an aromatase inhibitor with the presence of vaginal dryness or dyspareunia of sufficient severity to make the subject patient desire therapeutic intervention
* Vaginal dryness or dyspareunia must be present for at least two months prior to study entry
* Subjects must be on current treatment with tamoxifen or an aromatase inhibitor for at least two months prior to study enrollment (defined as the date of consent) and should not be planning to discontinue treatment or to change dose or type of endocrine treatment during the duration of the study
* Subjects must agree to not use any over-the-counter or prescription vaginal preparations (lubricants, creams, gels, ointments, solutions) during the four weeks of treatment with topical fluocinonide cream
* Subjects must agree to not use any medications, products, or preparations known to contain estrogen during the four weeks of treatment with topical fluocinonide cream
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Subjects must have ability to read, comprehend, and complete patient questionnaires independently or with assistance
* Subjects must sign informed consent
* Subjects must agree to read patient instructions regarding use of barrier contraceptive devices while on treatment with fluocinonide cream in the informed consent

Exclusion Criteria:

* Use of any vaginal preparations within one week prior to study enrollment (exception: subjects currently using a vaginal preparation can enroll after discontinuing treatment for 7 days)
* Use of any estrogen containing medications, products, or preparations
* Use of any systemic oral or parenteral steroid containing medications is not permitted; use of "High Daily Dose" inhaled/intranasal corticosteroids is not permitted; use inhaled/intranasal corticosteroid preparations at dosing levels less than "High Daily Dose" is permitted
* Current or past treatment with fluocinonide cream for vaginal dryness, itching, or dyspareunia
* Subject reported symptoms of vaginal infection with significant vaginal discharge or odor
* Known current vaginal infection
* Known vaginal pathology other than vaginal atrophy that could explain vaginal symptoms
* Known intolerance of topical steroid preparations
* Pregnant or lactating women (to be obtained via subject report only)
* Known diagnoses of diabetes mellitus, adrenal insufficiency (Addison's disease), or Cushing's syndrome
* No prior chemotherapeutic treatment for any malignancy other than breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Kemmer, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Supportive Care (Fluocinonide Cream): This is a single-arm, single-stage, open-label phase II trial of topical fluocinonide 0.05% cream to improve vaginal symptoms.
  All subjects will receive topical fluocinonide 0.05% cream to apply twice daily for two weeks and then once daily for two weeks to the vagina. The duration of treatment will be 4 weeks.
Period: Overall Study
Arm/Group | Supportive Care (Fluocinonide Cream)
Started | 34
Completed | 30
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: An intent-to-treat analysis set will include those who are enrolled in the trial regardless of the number of treatments received. All primary analyses will be conducted using the intent-to-treat analysis set. A safety analysis set will include those who receive at least one treatment.
Groups:
- Supportive Care: This is a single-arm, single-stage, open-label phase II trial of topical fluocinonide 0.05% cream to improve vaginal symptoms.
  All subjects will receive topical fluocinonide 0.05% cream to apply twice daily for two weeks and then once daily for two weeks to the vagina. The duration of treatment will be 4 weeks.
Arm/Group | Supportive Care
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.44 (9.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 0
Menopause status [Count of Participants; unit: Participants] — Pre-menopausal versus post-menopausal (defined as either no menses ≥ 12 months, medical ovarian suppression with leuprolide or goserelin, bilateral ovarian ablation with radiation, or bilateral oophorectomy)
  The subject's menopausal status will be classified according to the menopausal status at the time of enrollment on study.
  Participants
    Pre-menopausal | 1
    Post-menopausal | 33
Current endocrine therapy [Count of Participants; unit: Participants] — type of endocrine therapy currently taken by the subject
  tamoxifen vs. anastrazole vs. letrozole vs. exemestane
  Participants
    Anastrazole | 7
    Exemestane | 3
    Letrozole | 13
    Tamoxifen | 11
Prior cytotoxic chemotherapy received [Count of Participants; unit: Participants] — Whether the subject has received prior cytotoxic chemotherapy for breast cancer: prior cytotoxic chemotherapy versus no prior cytotoxic chemotherapy for breast cancer
  Participants
    Prior cytotoxic chemotherapy | 14
    No prior cytotoxic chemotherapy | 20
Indications for endocrine therapy [Count of Participants; unit: Participants] — use of endocrine therapy for preventative treatment with an increased risk for breast cancer vs. adjuvant treatment for a history of invasive breast cancer
  Participants
    Adjuvant | 33
    Prophylaxis | 1
Severe baseline symptoms, Dryness [Count of Participants; unit: Participants] — Severe symptoms indicated by a score of 3 or 4. Measured at study baseline
  Participants
    Severe | 15
    Not severe | 19
Severe baseline symptoms, Dyspareunia [Count of Participants; unit: Participants] — Severe symptoms indicated by a score of 3 or 4. Measured at study baseline
  Participants
    Severe | 15
    Not severe | 10
    Missing/not reported | 9
Severe baseline symptoms, Itching [Count of Participants; unit: Participants] — Severe symptoms indicated by a score of 3 or 4. Measured at study baseline
  Participants
    Severe | 1
    Not severe | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Symptom Scores of Vaginal Dryness
Description: Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively). Analyzed using Wilcoxon signed rank test with 2.5% significance level to account for two co-primary endpoints.
  Outcome measures median change in score from baseline to end of study. Scale is explained above for the scoring of symptoms at each time point. The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
Time Frame: Baseline and 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale | -2 [-3 to -1]
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); The primary endpoints (i.e., change in symptoms of vaginal dryness from the baseline to 4 weeks, and change in symptoms of dyspareunia from the baseline to 4 weeks) will be analyzed using Wilcoxon signed rank test with 2.5% significance level to account for two co-primary endpoints; Test type: Other — Two-sided test that the change is different from zero. Not tested against alternative treatment; single arm study; p < 0.001, Wilcoxon (Mann-Whitney) — 2.5% significance level to account for two co-primary endpoints
Statistical Analysis 2: Comparison: Supportive Care (Fluocinonide Cream); GEE (general estimating equation) methods were planned as a secondary analysis of the primary endpoints. Missing data for some of the weeks prevented these models from converging and we could not obtain valid results with these methods. Since this is a secondary analysis, we decided to compare symptom severity at baseline vs. week 4 (end of study). Symptoms are considered "severe" for scores 3 or 4 and "not severe" for scores 0, 1, 2; Test type: Other — Exact McNemar's test was used to test if the proportion of severe symptoms at baseline are equal to the proportion of severe symptoms at the end of the study; p = 0.001, McNemar — Since there are two-co-primary endpoints, the significance level is 2.5%; Odds Ratio (OR) = 0, 95% CI 2-sided [0 to 0.36]

2. Primary Outcome: Change in Symptom Scores of Dyspareunia
Description: as for outcome 1
Time Frame: Baseline and 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale | -2 [-3 to -1.8]
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); [analysis description as in outcome 1, analysis 1]; Test type: Other — Two-sided test that the change is different from zero. Not tested against alternative treatment; single arm study; p = 0.002, Wilcoxon (Mann-Whitney) — 2.5% significance level to account for two co-primary endpoints
Statistical Analysis 2: Comparison: Supportive Care (Fluocinonide Cream); GEE (general estimating equations) methods were planned as a secondary analysis of the primary endpoints. Missing data for some of the weeks prevented these models from converging and we could not obtain valid results with these methods. Since this is a secondary analysis, we decided to compare symptom severity at baseline vs. week 4 (end of study). Symptoms are considered "severe" for scores 3 or 4 and "not severe" for scores 0, 1, 2; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.062, McNemar — Since there are two-co-primary endpoints, the significance level is 2.5%; Odds Ratio (OR) = 0, 95% CI 2-sided [0 to 1.09]

3. Secondary Outcome: Change in Symptom Scores of Vaginal Itching
Description: Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively). Analyzed using Wilcoxon signed rank test with 2.5% significance level to account for two co-secondary endpoints.
  Outcome measures median change in score from baseline to end of study. Scale is explained above for the scoring of symptoms at each time point. The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
Time Frame: Baseline and 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale | -1 [-2 to 0]
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); The secondary endpoints (i.e., change in symptoms of vaginal itching from the baseline to 4 weeks, and change in vaginal index score from the baseline to 4 weeks) will be analyzed using Wilcoxon signed rank test with 2.5% significance level to account for two co-secondary endpoints; Test type: Other — Two-sided test that the change is different from zero. Not tested against alternative treatment; single arm study; p = 0.001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Total Vaginal Index Score.
Description: Change in total vaginal index score. The total vaginal index score is a numerical value ranging from zero to twelve, comprised of the three components of vaginal dryness, vaginal itching, and dyspareunia graded on an ordinal scale of zero to four added together.
  Outcome measures median change in score from baseline to end of study. Scale is explained above for the scoring of symptoms at each time point. The median change (i.e. median difference) can range from -12 to +12; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
  Analyzed using Wilcoxon signed rank test with 2.5% significance level to account for two co-secondary endpoints.
Time Frame: Baseline and 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale | -5 [-6 to -3.8]
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); [analysis description as in outcome 3, analysis 1]; Test type: Other — 2.5% significance level to account for two co-primary endpoints; p = 0.002, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Patients Experiencing Toxicities
Description: Toxicity data will be reported as descriptive data as the percentage of patients experiencing reported side effects. Toxicity and safety analyses will be conducted using the safety analysis set.
Time Frame: Over 4 weeks
Population: Toxicity and safety analyses will be conducted using the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
Participants | 1

6. Secondary Outcome: Change in Vaginal Dryness Symptom Scores by Age Characteristics
Description: Association of response in symptoms with characteristics of the subject population (Dryness and Age)
  Determine if there is an association between response in symptoms of vaginal dryness, itching, and/or dyspareunia with characteristics of the subject population.
  Response in symptoms is calculated as change in symptom score from baseline to week 4 (end of study). Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively).The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
Time Frame: Baseline and 4 weeks
Population: The rows are sub-groups of the total number analyzed. The sum of the row counts matches the overall number.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale
  Age 18-45: number analyzed (Participants) | 6
  Age 18-45 | -1.5 [-2.5 to -1.0]
  Age 46-55: number analyzed (Participants) | 10
  Age 46-55 | -2.0 [-3.0 to -2.0]
  Age 56-65: number analyzed (Participants) | 13
  Age 56-65 | -2.0 [-2.0 to -1.5]
  Age > 65: number analyzed (Participants) | 5
  Age > 65 | -2.0 [-3.0 to -0.75]
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); In order to compare the response between groups, Kruskal-Wallis ANOVA was used; Test type: Other; p = 0.1029, ANOVA — No adjustment for multiple comparison. Significance level of 0.05. Since this endpoint is of an exploratory nature and the significance is well above the threshold, not much more consideration was given to the issue of multiple comparisons; Kruskal-Wallis ANOVA rather than ANOVA since normal distribution of residuals may be suspect

7. Secondary Outcome: Change in Dyspareunia Symptom Scores by Age Characteristics
Description: Association of response in symptoms with characteristics of the subject population (Dyspareunia and Age)
  Determine if there is an association between response in symptoms of vaginal dryness, itching, and/or dyspareunia with characteristics of the subject population.
  Response in symptoms is calculated as change in symptom score from baseline to week 4 (end of study). Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively).The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
Time Frame: Baseline and 4 weeks
Population: The rows are sub-groups of the total number analyzed. The sum of the row counts matches the overall number.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale
  Age 18-45: number analyzed (Participants) | 6
  Age 18-45 | -1 [-1 to -1]
  Age 46-55: number analyzed (Participants) | 10
  Age 46-55 | -2 [-2 to -2]
  Age 56-65: number analyzed (Participants) | 13
  Age 56-65 | -2.5 [-3 to -1.75]
  Age > 65: number analyzed (Participants) | 5
  Age > 65 | -3 [-3 to -3]
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); In order to compare the response between groups, Kruskal-Wallis ANOVA was used; Test type: Other; p = 0.2678, ANOVA — [p-value comment as in outcome 6, analysis 1]; Kruskal-Wallis ANOVA rather than ANOVA since normal distribution of residuals may be suspect

8. Secondary Outcome: Change in Vaginal Itching Symptom Scores by Age Characteristics
Description: Association of response in symptoms with characteristics of the subject population (Itching and Age)
  Determine if there is an association between response in symptoms of vaginal dryness, itching, and/or dyspareunia with characteristics of the subject population.
  Response in symptoms is calculated as change in symptom score from baseline to week 4 (end of study). Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively).The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
Time Frame: Baseline and 4 weeks
Population: The rows are sub-groups of the total number analyzed. The sum of the row counts matches the overall number.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale
  Age 18-45: number analyzed (Participants) | 6
  Age 18-45 | -0.5 [-1.25 to 0.25]
  Age 46-55: number analyzed (Participants) | 10
  Age 46-55 | -1 [-2 to 0]
  Age 56-65: number analyzed (Participants) | 13
  Age 56-65 | -1 [-1.75 to 0]
  Age > 65: number analyzed (Participants) | 5
  Age > 65 | -0.5 [-1.25 to 0]
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); In order to compare the response between groups, Kruskal-Wallis ANOVA was used; Test type: Other; p = 0.2472, ANOVA — [p-value comment as in outcome 6, analysis 1]; Kruskal-Wallis ANOVA rather than ANOVA since normal distribution of residuals may be suspect

9. Secondary Outcome: Change in Vaginal Dryness Symptom Scores by Menopause Status Characteristics
Description: Association of response in symptoms with characteristics of the subject population (Dryness and Menopause status)
  Determine if there is an association between response in symptoms of vaginal dryness, itching, and/or dyspareunia with characteristics of the subject population.
  Response in symptoms is calculated as change in symptom score from baseline to week 4 (end of study). Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively).The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
Time Frame: Baseline and 4 weeks
Population: The rows are sub-groups of the total number analyzed. The sum of the row counts matches the overall number.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale
  Pre-Menopause: number analyzed (Participants) | 1
  Pre-Menopause | -2 [-2 to -2]
  Post-menopause: number analyzed (Participants) | 33
  Post-menopause | -2 [-3 to -1]
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); In order to compare the response between groups, Kruskal-Wallis ANOVA was used; Test type: Other; p = 0.507, ANOVA — [p-value comment as in outcome 6, analysis 1]; Kruskal-Wallis ANOVA rather than ANOVA since normal distribution of residuals may be suspect

10. Secondary Outcome: Change in Dyspareunia Symptom Scores by Menopause Status Characteristics
Description: Association of response in symptoms with characteristics of the subject population (Dyspareunia and Menopause status)
  Determine if there is an association between response in symptoms of vaginal dryness, itching, and/or dyspareunia with characteristics of the subject population.
  Response in symptoms is calculated as change in symptom score from baseline to week 4 (end of study). Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively).The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
Time Frame: Baseline and 4 weeks
Population: The rows are sub-groups of the total number analyzed. The sum of the row counts matches the overall number.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale
  Pre-Menopause: number analyzed (Participants) | 1
  Pre-Menopause | NA [NA to NA] — Missing data for the one subject in this group.
  Post-menopause: number analyzed (Participants) | 33
  Post-menopause | -2 [-3 to -1.75]
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); In order to compare the response between groups, Kruskal-Wallis ANOVA was used; Test type: Other; p = 0.3676, ANOVA — [p-value comment as in outcome 6, analysis 1]; Kruskal-Wallis ANOVA rather than ANOVA since normal distribution of residuals may be suspect

11. Secondary Outcome: Change in Vaginal Itching Symptom Scores by Menopause Status Characteristics
Description: Association of response in symptoms with characteristics of the subject population (Itching and Menopause status)
  Determine if there is an association between response in symptoms of vaginal dryness, itching, and/or dyspareunia with characteristics of the subject population.
  Response in symptoms is calculated as change in symptom score from baseline to week 4 (end of study). Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively).The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
Time Frame: Baseline and 4 weeks
Population: The rows are sub-groups of the total number analyzed. The sum of the row counts matches the overall number.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale
  Pre-Menopause: number analyzed (Participants) | 1
  Pre-Menopause | -1 [-1 to -1]
  Post-menopause: number analyzed (Participants) | 33
  Post-menopause | -1 [-2 to 0]
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); In order to compare the response between groups, Kruskal-Wallis ANOVA was used; Test type: Other; p = 0.6023, ANOVA — [p-value comment as in outcome 6, analysis 1]; Kruskal-Wallis ANOVA rather than ANOVA since normal distribution of residuals may be suspect

12. Secondary Outcome: Change in Vaginal Dryness Symptom Scores by Current Endocrine Therapy Characteristics
Description: Association of response in symptoms with characteristics of the subject population (Dryness and current endocrine therapy)
  Determine if there is an association between response in symptoms of vaginal dryness, itching, and/or dyspareunia with characteristics of the subject population.
  Response in symptoms is calculated as change in symptom score from baseline to week 4 (end of study). Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively).The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
Time Frame: Baseline and 4 weeks
Population: The rows are sub-groups of the total number analyzed. The sum of the row counts matches the overall number.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale
  Anastrazole: number analyzed (Participants) | 7
  Anastrazole | -2 [-2.75 to -2.0]
  Exemestane: number analyzed (Participants) | 3
  Exemestane | -2 [-2.5 to -1.5]
  Letrozole: number analyzed (Participants) | 13
  Letrozole | -2 [-3 to -1]
  Tamoxifen: number analyzed (Participants) | 11
  Tamoxifen | -2 [-2 to -1.25]
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); In order to compare the response between groups, Kruskal-Wallis ANOVA was used; Test type: Other; p = 0.6587, ANOVA — [p-value comment as in outcome 6, analysis 1]; Kruskal-Wallis ANOVA rather than ANOVA since normal distribution of residuals may be suspect

13. Secondary Outcome: Change in Dyspareunia Symptom Scores by Current Endocrine Therapy Characteristics
Description: Association of response in symptoms with characteristics of the subject population (Dyspareunia and current endocrine therapy)
  Determine if there is an association between response in symptoms of vaginal dryness, itching, and/or dyspareunia with characteristics of the subject population.
  Response in symptoms is calculated as change in symptom score from baseline to week 4 (end of study). Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively).The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
Time Frame: Baseline and 4 weeks
Population: The rows are sub-groups of the total number analyzed. The sum of the row counts matches the overall number.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale
  Anastrazole: number analyzed (Participants) | 7
  Anastrazole | -2 [-2.5 to -1.5]
  Exemestane: number analyzed (Participants) | 3
  Exemestane | -2 [-2 to -2]
  Letrozole: number analyzed (Participants) | 13
  Letrozole | -2.5 [-3 to -2]
  Tamoxifen: number analyzed (Participants) | 11
  Tamoxifen | -1.5 [-1.75 to -1.25]
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); In order to compare the response between groups, Kruskal-Wallis ANOVA was used; Test type: Other; p = 0.8772, ANOVA — [p-value comment as in outcome 6, analysis 1]; Kruskal-Wallis ANOVA rather than ANOVA since normal distribution of residuals may be suspect

14. Secondary Outcome: Change in Vaginal Itching Symptom Scores by Current Endocrine Therapy Characteristics
Description: Association of response in symptoms with characteristics of the subject population (Itching and current endocrine therapy)
  Determine if there is an association between response in symptoms of vaginal dryness, itching, and/or dyspareunia with characteristics of the subject population.
  Response in symptoms is calculated as change in symptom score from baseline to week 4 (end of study). Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively).The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
Time Frame: Baseline and 4 weeks
Population: The rows are sub-groups of the total number analyzed. The sum of the row counts matches the overall number.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale
  Anastrazole: number analyzed (Participants) | 7
  Anastrazole | -0.5 [-1 to 0]
  Exemestane: number analyzed (Participants) | 3
  Exemestane | -1 [-1.5 to -0.5]
  Letrozole: number analyzed (Participants) | 13
  Letrozole | -0.5 [-2 to 0]
  Tamoxifen: number analyzed (Participants) | 11
  Tamoxifen | -1 [-1.75 to -1]
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); In order to compare the response between groups, Kruskal-Wallis ANOVA was used; Test type: Other; p = 0.7395, ANOVA — [p-value comment as in outcome 6, analysis 1]; Kruskal-Wallis ANOVA rather than ANOVA since normal distribution of residuals may be suspect

15. Secondary Outcome: Change in Vaginal Dryness Symptom Scores by Prior Cytotoxic Therapy Characteristics
Description: Association of response in symptoms with characteristics of the subject population (Dryness and prior cytotoxic therapy)
  Determine if there is an association between response in symptoms of vaginal dryness, itching, and/or dyspareunia with characteristics of the subject population.
  Response in symptoms is calculated as change in symptom score from baseline to week 4 (end of study). Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively).The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
Time Frame: Baseline and 4 weeks
Population: The rows are sub-groups of the total number analyzed. The sum of the row counts matches the overall number.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale
  Yes: number analyzed (Participants) | 14
  Yes | -2 [-2 to -1]
  No: number analyzed (Participants) | 20
  No | -2 [-3 to -1]
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); In order to compare the response between groups, Kruskal-Wallis ANOVA was used; Test type: Other; p = 0.9618, ANOVA — [p-value comment as in outcome 6, analysis 1]; Kruskal-Wallis ANOVA rather than ANOVA since normal distribution of residuals may be suspect

16. Secondary Outcome: Change in Dyspareunia Symptom Scores by Prior Cytotoxic Therapy Characteristics
Description: Association of response in symptoms with characteristics of the subject population (Dyspareunia and prior cytotoxic therapy)
  Determine if there is an association between response in symptoms of vaginal dryness, itching, and/or dyspareunia with characteristics of the subject population.
  Response in symptoms is calculated as change in symptom score from baseline to week 4 (end of study). Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively).The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
Time Frame: Baseline and 4 weeks
Population: The rows are sub-groups of the total number analyzed. The sum of the row counts matches the overall number.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale
  Yes: number analyzed (Participants) | 14
  Yes | -2 [-2.25 to -1]
  No: number analyzed (Participants) | 20
  No | -2.5 [-3 to -2]
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); In order to compare the response between groups, Kruskal-Wallis ANOVA was used; Test type: Other; p = 0.5113, ANOVA — [p-value comment as in outcome 6, analysis 1]; Kruskal-Wallis ANOVA rather than ANOVA since normal distribution of residuals may be suspect

17. Secondary Outcome: Change in Vaginal Itching Symptom Scores by Prior Cytotoxic Therapy Characteristics
Description: Association of response in symptoms with characteristics of the subject population (Itching and prior cytotoxic therapy)
  Determine if there is an association between response in symptoms of vaginal dryness, itching, and/or dyspareunia with characteristics of the subject population.
  Response in symptoms is calculated as change in symptom score from baseline to week 4 (end of study). Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively).The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
Time Frame: Baseline and 4 weeks
Population: The rows are sub-groups of the total number analyzed. The sum of the row counts matches the overall number.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale
  Yes: number analyzed (Participants) | 14
  Yes | -1 [-1 to 0]
  No: number analyzed (Participants) | 20
  No | -1 [-2 to 0]
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); In order to compare the response between groups, Kruskal-Wallis ANOVA was used; Test type: Other; p = 0.8833, ANOVA — [p-value comment as in outcome 6, analysis 1]; Kruskal-Wallis ANOVA rather than ANOVA since normal distribution of residuals may be suspect

18. Secondary Outcome: Change in Vaginal Dryness Symptom Scores by Indication for Endocrine Therapy Characteristics
Description: Association of response in symptoms with characteristics of the subject population (Dryness and Indications)
  Determine if there is an association between response in symptoms of vaginal dryness, itching, and/or dyspareunia with characteristics of the subject population.
  Response in symptoms is calculated as change in symptom score from baseline to week 4 (end of study). Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively).The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
Time Frame: Baseline and 4 weeks
Population: The rows are sub-groups of the total number analyzed. The sum of the row counts matches the overall number.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale
  Adjuvant: number analyzed (Participants) | 33
  Adjuvant | -2 [-2.5 to -1]
  Prophylaxis: number analyzed (Participants) | 1
  Prophylaxis | -3 [-3 to -3]
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); In order to compare the response between groups, Kruskal-Wallis ANOVA was used; Test type: Other; p = 0.7983, ANOVA — [p-value comment as in outcome 6, analysis 1]; Kruskal-Wallis ANOVA rather than ANOVA since normal distribution of residuals may be suspect

19. Secondary Outcome: Change in Dyspareunia Symptom Scores by Indication for Endocrine Therapy Characteristics
Description: Association of response in symptoms with characteristics of the subject population (Dyspareunia and Indications)
  Determine if there is an association between response in symptoms of vaginal dryness, itching, and/or dyspareunia with characteristics of the subject population.
  Response in symptoms is calculated as change in symptom score from baseline to week 4 (end of study). Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively).The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
Time Frame: Baseline and 4 weeks
Population: The rows are sub-groups of the total number analyzed. The sum of the row counts matches the overall number.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale
  Adjuvant: number analyzed (Participants) | 33
  Adjuvant | -2 [-3 to -1.75]
  Prophylaxis: number analyzed (Participants) | 1
  Prophylaxis | NA [NA to NA] — Data for single participant is missing
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); In order to compare the response between groups, Kruskal-Wallis ANOVA was used; Test type: Other; p = 0.4937, ANOVA — [p-value comment as in outcome 6, analysis 1]; Kruskal-Wallis ANOVA rather than ANOVA since normal distribution of residuals may be suspect

20. Secondary Outcome: Change in Vaginal Itching Symptom Scores by Indication for Endocrine Therapy Characteristics
Description: Association of response in symptoms with characteristics of the subject population (Itching and Indications)
  Determine if there is an association between response in symptoms of vaginal dryness, itching, and/or dyspareunia with characteristics of the subject population.
  Response in symptoms is calculated as change in symptom score from baseline to week 4 (end of study). Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively).The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
Time Frame: Baseline and 4 weeks
Population: The rows are sub-groups of the total number analyzed. The sum of the row counts matches the overall number.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale
  Adjuvant: number analyzed (Participants) | 33
  Adjuvant | -1 [-1.75 to 0]
  Prophylaxis: number analyzed (Participants) | 1
  Prophylaxis | -2 [-2 to -2]
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); In order to compare the response between groups, Kruskal-Wallis ANOVA was used; Test type: Other; p = 0.9106, ANOVA — [p-value comment as in outcome 6, analysis 1]; Kruskal-Wallis ANOVA rather than ANOVA since normal distribution of residuals may be suspect

21. Secondary Outcome: Change in Vaginal Dryness Symptom Scores by Patient Reported Compliance Characteristics
Description: Association of response in symptoms with patient reported compliance (Dryness)
  Determine if there is an association between response in symptoms of vaginal dryness, itching, and/or dyspareunia with patient reported compliance.
  Response in symptoms is calculated as change in symptom score from baseline to week 4 (end of study). Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively).The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
  Groups are made by % of compliance reported by patients
Time Frame: Baseline and 4 weeks
Population: The rows are sub-groups of the total number analyzed. The sum of the row counts matches the overall number.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale
  50 - 74%: number analyzed (Participants) | 1
  50 - 74% | -2 [-2 to -2]
  >= 75%: number analyzed (Participants) | 29
  >= 75% | -2 [-3 to -1]
  Missing / not reported: number analyzed (Participants) | 4
  Missing / not reported | NA [NA to NA] — Data is missing for these patients
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); In order to compare the response between groups, Kruskal-Wallis ANOVA was used; Test type: Other; p = 0.507, ANOVA — [p-value comment as in outcome 6, analysis 1]; Kruskal-Wallis ANOVA rather than ANOVA since normal distribution of residuals may be suspect

22. Secondary Outcome: Change in Dyspareunia Symptom Scores by Patient Reported Compliance Characteristics
Description: Association of response in symptoms with patient reported compliance (Dyspareunia)
  Determine if there is an association between response in symptoms of vaginal dryness, itching, and/or dyspareunia with patient reported compliance.
  Response in symptoms is calculated as change in symptom score from baseline to week 4 (end of study). Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively).The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
  Groups are made by % of compliance reported by patients
Time Frame: Baseline and 4 weeks
Population: The rows are sub-groups of the total number analyzed. The sum of the row counts matches the overall number.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale
  50 - 74%: number analyzed (Participants) | 1
  50 - 74% | NA [NA to NA] — Data is missing; could not calculate
  >= 75%: number analyzed (Participants) | 29
  >= 75% | -2 [-3 to -1.75]
  Missing / not reported: number analyzed (Participants) | 4
  Missing / not reported | NA [NA to NA] — Data is missing; could not calculate
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); In order to compare the response between groups, Kruskal-Wallis ANOVA was used; Test type: Other; p = 0.3676, ANOVA — [p-value comment as in outcome 6, analysis 1]; Kruskal-Wallis ANOVA rather than ANOVA since normal distribution of residuals may be suspect

23. Secondary Outcome: Change in Vaginal Itching Symptom Scores by Patient Reported Compliance Characteristics
Description: Association of response in symptoms with patient reported compliance (Itching)
  Determine if there is an association between response in symptoms of vaginal dryness, itching, and/or dyspareunia with patient reported compliance.
  Response in symptoms is calculated as change in symptom score from baseline to week 4 (end of study). Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively).The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
  Groups are made by % of compliance reported by patients
Time Frame: Baseline and 4 weeks
Population: The rows are sub-groups of the total number analyzed. The sum of the row counts matches the overall number.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale
  50 - 74%: number analyzed (Participants) | 1
  50 - 74% | -1 [-1 to -1]
  >= 75%: number analyzed (Participants) | 29
  >= 75% | -1 [-2 to 0]
  Missing / not reported: number analyzed (Participants) | 4
  Missing / not reported | NA [NA to NA] — Data is missing; could not calculate.
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); In order to compare the response between groups, Kruskal-Wallis ANOVA was used; Test type: Other; p = 0.6023, ANOVA — [p-value comment as in outcome 6, analysis 1]; Kruskal-Wallis ANOVA rather than ANOVA since normal distribution of residuals may be suspect

24. Secondary Outcome: Change in Vaginal Dryness Symptom Scores by Tube Weight Based Compliance Characteristics
Description: Association of response in symptoms with tube weight based compliance (Dryness)
  Determine if there is an association between response in symptoms of vaginal dryness, itching, and/or dyspareunia with compliance determined by % of tube used by weight.
  Response in symptoms is calculated as change in symptom score from baseline to week 4 (end of study). Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively).The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
  Groups are made by % of tube used by weight.
Time Frame: Baseline and 4 weeks
Population: The rows are sub-groups of the total number analyzed. The sum of the row counts matches the overall number.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale
  < 25%: number analyzed (Participants) | 5
  < 25% | -1 [-1 to -1]
  25 - 49%: number analyzed (Participants) | 8
  25 - 49% | -2 [-3 to -1.75]
  50 - 74%: number analyzed (Participants) | 8
  50 - 74% | -2 [-3 to -1.75]
  >= 75%: number analyzed (Participants) | 7
  >= 75% | -2 [-2 to -2]
  Missing / not reported: number analyzed (Participants) | 6
  Missing / not reported | -2.5 [-3.25 to -1.75]
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); In order to compare the response between groups, Kruskal-Wallis ANOVA was used; Test type: Other; p = 0.08531, ANOVA — [p-value comment as in outcome 6, analysis 1]; Kruskal-Wallis ANOVA rather than ANOVA since normal distribution of residuals may be suspect

25. Secondary Outcome: Change in Dyspareunia Symptom Scores by Tube Weight Based Compliance Characteristics
Description: Association of response in symptoms with tube weight based compliance (Dyspareunia)
  Determine if there is an association between response in symptoms of vaginal dryness, itching, and/or dyspareunia with compliance determined by % of tube used by weight.
  Response in symptoms is calculated as change in symptom score from baseline to week 4 (end of study). Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively).The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
  Groups are made by % of tube used by weight.
Time Frame: Baseline and 4 weeks
Population: The rows are sub-groups of the total number analyzed. The sum of the row counts matches the overall number.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale
  < 25%: number analyzed (Participants) | 5
  < 25% | -1 [-1 to -1]
  25 - 49%: number analyzed (Participants) | 8
  25 - 49% | -2 [-2.5 to -1.5]
  50 - 74%: number analyzed (Participants) | 8
  50 - 74% | -2 [-2.25 to -1.75]
  >= 75%: number analyzed (Participants) | 7
  >= 75% | -2 [-2.25 to -2]
  Missing / not reported: number analyzed (Participants) | 6
  Missing / not reported | -3 [-3 to -3]
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); In order to compare the response between groups, Kruskal-Wallis ANOVA was used; Test type: Other; p = 0.2011, ANOVA — [p-value comment as in outcome 6, analysis 1]; Kruskal-Wallis ANOVA rather than ANOVA since normal distribution of residuals may be suspect

26. Secondary Outcome: Change in Vaginal Itching Symptom Scores by Tube Weight Based Compliance Characteristics
Description: Association of response in symptoms with tube weight based compliance (Itching)
  Determine if there is an association between response in symptoms of vaginal dryness, itching, and/or dyspareunia with compliance determined by % of tube used by weight.
  Response in symptoms is calculated as change in symptom score from baseline to week 4 (end of study). Change in symptom scores of vaginal dryness, itching, and dyspareunia will be evaluated by the Mayo/North Central Cancer Treatment Group (NCCTG) patient questionnaire which has patients grade how much vaginal dryness, vaginal itching, and vaginal discomfort during intercourse they are currently experiencing on an ordinal scale of zero to four (none, mild, moderate, severe, and very severe, respectively).The median change (i.e. median difference) can range from -4 to +4; negative values indicate improved symptoms, zero no change, and positive values indicate worsened symptoms.
  Groups are made by % of tube used by weight.
Time Frame: Baseline and 4 weeks
Population: The rows are sub-groups of the total number analyzed. The sum of the row counts matches the overall number.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Supportive Care (Fluocinonide Cream)
Number analyzed (Participants) | 34
units on a scale
  < 25%: number analyzed (Participants) | 5
  < 25% | -1 [-1 to -1]
  25 - 49%: number analyzed (Participants) | 8
  25 - 49% | -1 [-2 to 0]
  50 - 74%: number analyzed (Participants) | 8
  50 - 74% | 0 [-1 to 0]
  >= 75%: number analyzed (Participants) | 7
  >= 75% | -1 [-2 to -0.5]
  Missing / not reported: number analyzed (Participants) | 6
  Missing / not reported | -1 [-1.5 to -0.5]
Statistical Analysis 1: Comparison: Supportive Care (Fluocinonide Cream); In order to compare the response between groups, Kruskal-Wallis ANOVA was used; Test type: Other; p = 0.1187, ANOVA — [p-value comment as in outcome 6, analysis 1]; Kruskal-Wallis ANOVA rather than ANOVA since normal distribution of residuals may be suspect

ADVERSE EVENTS:
Time Frame: End of study week 1, 2, 3, 4
Description: Toxicities and adverse events will be assessed using the NCI Common Toxicity Criteria (CTC) Version 4.0. Since CTEP has standardized the CTC, the NCI does not require the inclusion of the CTC within the protocol document. A copy can be downloaded from the CTEP home page (http://ctep.info.nih.gov).
Arm/Group | Supportive Care (Fluocinonide Cream)
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 24/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Fluocinonide Cream) (N=34)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 23 (23)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Vaginal discharge (Skin and subcutaneous tissue disorders) | 2 (2)
Vaginal inflammation (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Original plan was to use GEE modeling for secondary analysis of primary endpoints. Missing data and small counts caused us to perform this analysis using other statistical methods. Data was categorized and tested using McNemar's Test for results

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes